CLINICAL TRIAL: NCT02487797
Title: A Randomized Double Blind Clinical Trial Comparing Oxytocin Low-dose and High-dose Regimens for Labor Augmentation
Brief Title: Comparison of Low-dose and High-dose Oxytocin Regimens for Labor Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Moeun Son, Assistant Professor in Obstetrics and Gynecology - Maternal Fetal Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00201148
Record Dates: First submitted 2015-06-09; First posted 2015-07-01 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Dystocia
MeSH Terms: conditions — Dystocia | interventions — Oxytocin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose oxytocin regimen (Experimental): The oxytocin solution will be prepared using 90 units of oxytocin in 500 milliliters of normal saline (sodium chloride 0.9%). The oxytocin infusion will be initiated with a starting oxytocin concentration rate of 6 milliunits/minute (volume rate 2 milliliters/hour) that can be increased at increments of 6 milliunits/minute (volume rate 2 milliliters/hour) every 15-30 minutes until a labor pattern with uterine contractions every 2-3 minutes of moderate to strong intensity is established.
  Interventions: Drug: Oxytocin; Other: Sodium Chloride 0.9%
- Low dose oxytocin regimen (Active Comparator): The oxytocin solution will be prepared using 30 units of oxytocin in 500 milliliters of normal saline (sodium chloride 0.9%). The oxytocin infusion will be initiated with a starting oxytocin concentration rate of 2 milliunits/minute (volume rate 2 milliliters/hour) that can be increased at increments of 2 milliunits/minute (volume rate 2 milliliters/hour) every 15-30 minutes until a labor pattern with uterine contractions every 2-3 minutes of moderate to strong intensity is established.
  Interventions: Drug: Oxytocin; Other: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Pitocin
Other: Sodium Chloride 0.9%
  Other Names: Normal Saline

SUMMARY:
Oxytocin is a medication that is often used to strengthen contractions to overcome delayed labor progress. The primary aim of this study is to determine whether receiving a higher dose of oxytocin lowers the chance of needing a cesarean section when compared to a lower dose of oxytocin. Other aims include examining the relationship between dose of oxytocin regimen and length of labor, postpartum hemorrhage, intrauterine infection, umbilical cord gas, neonatal Apgar score <5 at 5 minutes, and need for neonatal intensive care.

DETAILED DESCRIPTION:
This randomized double blind clinical trial of consenting nulliparous women in spontaneous labor who require oxytocin for labor augmentation seeks to determine whether use of a high dose oxytocin regimen improves obstetric outcomes when compared with a low dose oxytocin regimen, in a manner that is safe for both mother and neonate.

This project will include 1002 women recruited from the obstetrical service at Prentice Women's Hospital. Women will be included if they are at least 36 weeks gestation, have a singleton pregnancy, and have been diagnosed with spontaneous labor or spontaneous rupture of membranes. Women will be exposed to oxytocin for the indication of labor augmentation at the discretion of their obstetric provider.

Women will be randomized with equal probability to intervention group using a fixed allocation procedure. To maintain a double blind design, the Prentice Women's Hospital pharmacy will carry out the randomization of oxytocin solutions according to the random assignment so that neither the women or their care providers nor the investigators will know the identity of the intervention assignment. The low-dose oxytocin regimen group will receive a starting oxytocin regimen concentration rate of 2 milliunits/minute that can be increased at increments of 2 milliunits/minute, as per the discretion of their obstetric provider. The high-dose oxytocin regimen group will receive a starting oxytocin regimen concentration rate of 6 milliunits/minute that can be increased at increments of 6 milliunits/minute, as per the discretion of their obstetric provider.

Once the women are enrolled, randomized, and in receipt of their assigned interventions, further clinical management will be left to the discretion of each woman's obstetric provider.

Prior to discharge from the hospital, baseline demographic and clinical data will be obtained via chart review.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed written consent
* Age 18-45 years
* Nulliparous
* Pregnant with a live singleton gestation that is equal to or greater than 36 weeks
* Diagnosed with at least 6 regular uterine contractions in an observation period of no more than 60 minutes and at least one of the following: spontaneous rupture of membranes, OR cervix greater than or equal to 3 centimeters dilated OR cervix at least 80% effaced.
* The participant's attending obstetric physician or midwife has determined that the participant needs administration of oxytocin infusion for labor augmentation. Labor augmentation will be defined as stimulation of uterine contractions when spontaneous contractions have failed to result in progressive cervical dilation of descent of fetus.

Exclusion Criteria:

* Women not meeting the above criteria
* History of prior cesarean section or uterine surgery
* Fetus in non-cephalic presentation
* Participant is undergoing labor induction (i.e. cervical ripening)
* Non-English speaking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1003 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moeun Son, MD, MSCI, Principal Investigator — Northwestern University; Alan Peaceman, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Derived] Son M, Roy A, Grobman WA, Miller ES, Dude A, Peaceman AM, Stetson B. Maximum Dose Rate of Intrapartum Oxytocin Infusion and Associated Obstetric and Perinatal Outcomes. Obstet Gynecol. 2023 Feb 1;141(2):379-386. doi: 10.1097/AOG.0000000000005058. Epub 2023 Jan 4. PMID 36649339
- [Derived] Son M, Roy A, Stetson BT, Grady NT, Vanecko MC, Bond N, Swanson K, Grobman WA, Miller ES, Peaceman AM. High-Dose Compared With Standard-Dose Oxytocin Regimens to Augment Labor in Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):991-998. doi: 10.1097/AOG.0000000000004399. PMID 33957657

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Oxytocin Regimen: The oxytocin solution will be prepared using 90 units of oxytocin in 500 milliliters of normal saline (sodium chloride 0.9%). The oxytocin infusion will be initiated with a starting oxytocin concentration rate of 6 milliunits/minute (volume rate 2 milliliters/hour) that can be increased at increments of 6 milliunits/minute (volume rate 2 milliliters/hour) every 15-30 minutes until a labor pattern with uterine contractions every 2-3 minutes of moderate to strong intensity is established.
  Oxytocin
  Sodium Chloride 0.9%
- Low Dose Oxytocin Regimen: The oxytocin solution will be prepared using 30 units of oxytocin in 500 milliliters of normal saline (sodium chloride 0.9%). The oxytocin infusion will be initiated with a starting oxytocin concentration rate of 2 milliunits/minute (volume rate 2 milliliters/hour) that can be increased at increments of 2 milliunits/minute (volume rate 2 milliliters/hour) every 15-30 minutes until a labor pattern with uterine contractions every 2-3 minutes of moderate to strong intensity is established.
  Oxytocin
  Sodium Chloride 0.9%
Period: Overall Study
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Started | 502 | 501
Completed | 502 | 501
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen | Total
Number analyzed (Participants) | 502 | 501 | 1003
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (4.4) | 31.7 (4.3) | 31.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 502 | 501 | 1003
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 332 | 342 | 674
  Black | 36 | 44 | 80
  Hispanic or Latina | 27 | 26 | 53
  Asian or Pacific Islander | 42 | 47 | 89
  Other, unknown, or more than one race | 65 | 42 | 107
Married or living with a partner [Count of Participants; unit: Participants] | 396 | 409 | 805
Insurance type [Count of Participants; unit: Participants]
  Commercial | 435 | 442 | 877
  Government | 66 | 59 | 125
  Uninsured | 1 | 0 | 1
Body mass index at trial entry [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Data missing for 6 participants
  kg/m^2
    number analyzed (Participants) | 498 | 499 | 997
    (all) | 28.8 [26.4 to 32.0] | 29.9 [26.9 to 32.8] | 29.2 [26.6 to 32.5]
Gestational or pre-gestational diabetes [Count of Participants; unit: Participants] | 12 | 15 | 27
Chronic hypertension [Count of Participants; unit: Participants] | 6 | 4 | 10
Hypertensive disorders of pregnancy [Count of Participants; unit: Participants] | 47 | 63 | 110
Group B Streptococcus carrier [Count of Participants; unit: Participants] — Population: Data missing for total of 25 participants
  Participants
    number analyzed (Participants) | 492 | 486 | 978
    (all) | 95 | 88 | 183
Gestational age at trial entry (weeks) [Mean (Standard Deviation); unit: weeks] | 39.1 (0.8) | 39.1 (0.7) | 39.1 (0.7)
Indication for trial entry [Count of Participants; unit: Participants]
  Labor with intact membranes | 236 | 241 | 477
  Spontaneous rupture of membranes | 266 | 260 | 526
Receipt of magnesium sulfate infusion [Count of Participants; unit: Participants] | 10 | 13 | 23
Neuraxial analgesia before trial entry [Count of Participants; unit: Participants] | 246 | 247 | 493
Amniotomy before trial entry [Count of Participants; unit: Participants] | 110 | 125 | 235
Female fetal sex [Count of Participants; unit: Participants] | 268 | 239 | 507
Neonatal birthweight [Median (Inter-Quartile Range); unit: grams] | 3325 [3070 to 3625] | 3350 [3080 to 3610] | 3335 [3080 to 3625]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Delivered by Cesarean
Description: Number of participants delivered by cesarean section
Time Frame: At time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 73 | 72

2. Secondary Outcome: Labor Augmentation Duration
Description: Time from randomization to delivery
Time Frame: Number of hours from randomization to delivery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
hours | 9.1 (5.6) | 10.5 (7.0)

3. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Description: Estimated blood loss greater than 500 milliliters after a vaginal delivery or greater than 1000 milliliters after a cesarean delivery
Time Frame: From date of delivery to date of hospital discharge, an expected average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 29 | 23

4. Secondary Outcome: Number of Participants With Intrapartum Chorioamnionitis
Description: Fever greater than 100.4 Fahrenheit in the intrapartum period with the initiation of a therapeutic antibiotic regimen in the intrapartum period
Time Frame: From time of labor admission to time of delivery, an expected average of 24 to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 52 | 78

5. Secondary Outcome: Number of Participants With Postpartum Endometritis
Description: Fever greater than 100.4 Fahrenheit in the postpartum period with the initiation of a therapeutic antibiotic regimen in the postpartum period
Time Frame: From time of delivery to time of hospital discharge, an expected average of 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 3 | 5

6. Secondary Outcome: Number of Participants Whose Offspring Experiences a Perinatal Death
Description: Perinatal death includes intrapartum stillbirth and neonatal death
Time Frame: Study enrollment to delivery (if intrapartum stillbirth) or 28 days of life (if liveborn)
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Umbilical Cord Acidemia
Description: Umbilical cord arterial blood pH less than 7.0 or base deficit greater than 12 mmol/L; or cord venous blood pH less than 7.0 or base deficit greater than 12 mmol/L when umbilical artery values are not available
Time Frame: At time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 14 | 27

8. Secondary Outcome: Neonatal Apgar Score of Less Than 3 at 5 Minutes of Life
Description: Number of participants with neonates with Apgar score of less than 3 at 5 minutes of life. This is using a Apgar scale which ranges from minimum total score of 0 and maximum total score of 10, with higher score representing a better outcome.
Time Frame: Delivery through 5 minutes of life
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 3 | 4

9. Secondary Outcome: Admission to Neonatal Intensive Care Unit
Description: Number of participants whose neonates are admitted to Neonatal Intensive Care Unit
Time Frame: Delivery to 28 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 29 | 33

10. Secondary Outcome: Number of Participants Whose Neonates Experience a Composite of Severe Neonatal Morbidity and Perinatal Mortality
Description: Neonatal composite morbidity will be defined as occurrence of any of the following: perinatal death, severe, respiratory distress, major birth injury, encephalopathy, seizure, need for hypothermic treatment, or sepsis
Time Frame: Delivery to 28 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
Number analyzed (Participants) | 502 | 501
Participants | 5 | 7

ADVERSE EVENTS:
Time Frame: Maternal adverse events were monitored from study enrollment until delivery hospitalization discharge, typically up to 5 days. Neonatal outcomes were monitored from birth until birth hospitalization discharge or 28 days of life, whichever came first.
Description: Unanticipated adverse events will be defined as any event that meets the following conditions: the event is not a known or reasonably foreseeable risk associated with the study procedures (e.g. risks related to administration of oxytocin and confidential information specified in the informed consent), and the event, in the investigators' opinion, is or could be directly related to the subject's participation in this research protocol.
Arm/Group | High Dose Oxytocin Regimen | Low Dose Oxytocin Regimen
All-Cause Mortality (participants affected / at risk) | 0/502 | 0/501
Serious Adverse Events (participants affected / at risk) | 0/502 | 0/501
Other Adverse Events (participants affected / at risk) | 0/502 | 0/501

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT02487797/Prot_SAP_000.pdf